CLINICAL TRIAL: NCT02711397
Title: Fecal Gluten Peptides Reveal Limitations of Serological Tests and Food Questionnaires for Monitoring Gluten-free Diet
Brief Title: Quantification of Gluten Peptides in Feces
Acronym: DELIAC
Status: Completed | Type: Observational
Sponsor: Biomedal S.L. (Other)
Responsible Party: Sponsor
Other Study IDs: DELIAC
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2016-03

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Celiac patients: Celiac patients following a GFD for at least one year prior to the inclusion in the study.
  Interventions: Other: Observational study
- Positive controls: Healthy children and adults on an unrestricted gluten containing diet.
  Interventions: Other: Observational study
- Negative controls: Healthy infants who were exclusively fed with infant formula specifically labelled as gluten-free.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Comparison excretion levels of gluten immunogenic peptides

SUMMARY:
Treatment for celiac disease (CD) is a lifelong strict gluten-free diet (GFD). Patients should be followed-up with dietary interviews and serologic tests for CD markers to ensure adherence to the diet. However, none of these methods offer an accurate measure of dietary compliance. Our aim was to evaluate the measurement of gluten immunogenic peptides (GIP) in stools as a marker of GFD adherence in CD patients and compare it with traditional methods of GFD monitoring.

We performed a prospective, non-randomized, multicentre study including 188 CD patients on a GFD and 73 healthy controls on a gluten-containing diet. Subjects were given a dietary questionnaire and fecal GIP quantified by ELISA (iVYLISA GIP-S kit). Serological anti-tissue transglutaminase (anti-tTG) IgA and anti-deamidated gliadin peptide (anti-DGP) IgA antibodies were measured simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* The study group consisted of celiac patients following a GFD for at least one year prior to the inclusion in the study and they were required to have an HLA-DQ2 or HLA-DQ8 haplotype and an histologically abnormal duodenal biopsy (grade Marsh IIIB or IIIC) at the time of diagnosis, supported by positive serum anti-endomysium IgA antibodies and/or anti-tissue transglutaminase (anti-tTG) IgA antibodies.
* The positive and negative control groups was comprised of healthy asymptomatic subjects in whom CD had been ruled out and who were not suspected of having any other gastrointestinal condition

Exclusion Criteria:

* All study patients included history of kidney or liver disease, and history of severe psychiatric disease or seizure disorder.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Celiac patients following a GFD for at least one year prior to the inclusion in the study
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Adherence to gluten-free diet | two years

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Sousa, PhD, Study Director — Department of Microbiology and Parasitology, Faculty of Pharmacy, University of Seville

REFERENCES:
- [Derived] Comino I, Segura V, Ortigosa L, Espin B, Castillejo G, Garrote JA, Sierra C, Millan A, Ribes-Koninckx C, Roman E, Rodriguez-Herrera A, Diaz J, Silvester JA, Cebolla A, Sousa C. Prospective longitudinal study: use of faecal gluten immunogenic peptides to monitor children diagnosed with coeliac disease during transition to a gluten-free diet. Aliment Pharmacol Ther. 2019 Jun;49(12):1484-1492. doi: 10.1111/apt.15277. Epub 2019 May 10. PMID 31074004
- [Derived] Comino I, Fernandez-Banares F, Esteve M, Ortigosa L, Castillejo G, Fambuena B, Ribes-Koninckx C, Sierra C, Rodriguez-Herrera A, Salazar JC, Caunedo A, Marugan-Miguelsanz JM, Garrote JA, Vivas S, Lo Iacono O, Nunez A, Vaquero L, Vegas AM, Crespo L, Fernandez-Salazar L, Arranz E, Jimenez-Garcia VA, Antonio Montes-Cano M, Espin B, Galera A, Valverde J, Giron FJ, Bolonio M, Millan A, Cerezo FM, Guajardo C, Alberto JR, Rosinach M, Segura V, Leon F, Marinich J, Munoz-Suano A, Romero-Gomez M, Cebolla A, Sousa C. Fecal Gluten Peptides Reveal Limitations of Serological Tests and Food Questionnaires for Monitoring Gluten-Free Diet in Celiac Disease Patients. Am J Gastroenterol. 2016 Oct;111(10):1456-1465. doi: 10.1038/ajg.2016.439. Epub 2016 Sep 20. PMID 27644734